CLINICAL TRIAL: NCT03519308
Title: A Pilot Study of Perioperative Nivolumab and Paricalcitol to Target the Microenvironment in Resectable Pancreatic Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The accrual goal could not be met and the drug manufacturer pulled support
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 22217
Record Dates: First submitted 2018-04-24; First posted 2018-05-08 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Nivolumab; 130-nm albumin-bound paclitaxel; Gemcitabine; paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Nivolumab; Drug: Nab-Paclitaxel; Drug: Gemcitabine; Drug: Paricalcitol
- Arm B (Experimental)
  Interventions: Drug: Nivolumab; Drug: Nab-Paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Nivolumab — Before Surgery Wks 1 &3, After Surgery Wks 1 &3
Drug: Nab-Paclitaxel — Wks 1,2,3 before surgery and Wks 1, 2,3 after surgery
Drug: Gemcitabine — Wks 1,2,3 before surgery and Wks 1,2,3 after surgery
Drug: Paricalcitol — Wks 1,2,3, 4 before surgery and Wks 1,2,3 after surgery
  Arms: Arm A

SUMMARY:
The main purpose of this study is to look at the potential effects of paricalcitol (a drug similar to vitamin D) and nivolumab on pancreatic tumors in patients who are treated with gemcitabine and abraxane. The study will also look at the safety of including paricalcitol and nivolumab as part of the gemcitabine and abraxane chemotherapeutic regimen.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, apparently resectable adenocarcinoma of the pancreas at registration.
* Age greater than or equal to 18 years
* ECOG performance status of 0-2.
* Standard laboratory criteria for hematologic, biochemical, and urinary indices within a range that, in the opinion of the physician, clinically supports enrollment of the subject on the trial.

  a. Note: subjects must have: Creatinine < 2xULN, Neutrophils >1.5x109/L, total bilirubin < 3xULN, AST <5xULN, ALT <5xULN, and Platelets >100,000/mm3
* Ability to provide written informed consent

Exclusion Criteria:

* Subjects with hypercalcemia (blood levels greater than 11.5 mg/dL). In subjects creatinine clearance <60mL/min, blood calcium levels must be 9.5 mg/dL or lower.
* Subjects who are currently pregnant, planning to become pregnant, or breast-feeding

  1. Females participants of child-bearing potential are required to use an effective contraception method (see Appendix A) or abstain from intercourse during treatment and for at least 5 months following the last dose
  2. Males participants with partners of child-bearing potential are required to use an effective contraception method (see Appendix A) or abstain from intercourse during treatment and for at least 5 months following the last dose 3. Subjects who, in the opinion of the physician, would not be clinically appropriate for receipt of the therapy regimen associated with participation 4. Subjects with contraindications to immune checkpoint therapy, as follows:

  <!-- -->

  1. Interstitial lung disease that is symptomatic or may interfere with the detection and management of suspected drug-related pulmonary toxicity
  2. Prior organ allograft or allogeneic bone marrow transplantation
  3. Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
  4. Active autoimmune disease, except for vitiligo, type 1 diabetes mellitus, asthma, atopic dermatitis, or endocrinopathies manageable by hormone replacement; other autoimmune conditions may be allowable at the discretion of the principal investigator
  5. Condition requiring systemic treatment with either corticosteroids

     * Systemic steroids at physiologic doses (equivalent to dose of oral prednisone 10 mg) are permitted. Steroids as anti-emetics for chemotherapy are strongly discouraged (see section 5.1.3)
     * Intranasal, inhaled, topical, intra-articular, and ocular corticosteroids with minimal systemic absorption are permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Dwyer, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment naïve patients with apparently resectable adenocarcinoma of the pancreas with the epithelial subtype were enrolled at the University of Pennsylvania from July 2020 through April 2022.
Pre-assignment Details: Patients pre-treated with chemotherapy nivolumab were randomized 1:1 to receive (Arm A) or not receive (Arm B) weekly intravenous paricalcitol. 3 patients were enrolled in the study, therefore, the target enrollment of 20 patients was not reached.
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with resectable epithelial-subtype pancreatic cancer
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Median (Full Range); unit: years] | 58.5 [56 to 61] | 57 [57 to 57] | 57 [56 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: An adverse event (AE) was defined as any unfavorable symptom, sign, illness or experience that occurs at any dose and develops or worsens in severity during the course of the study. AEs were graded using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Time Frame: 18 months
Population: participants
Measure: Mean (Standard Deviation); unit: number of adverse events
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 2 | 1
number of adverse events | 19 (4.2) | 27 (0)

2. Secondary Outcome: Objective Response Rate
Description: Objective response rate by RECIST v 1.1 after neoadjuvant chemotherapy. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 2 | 1
Participants | 1 | 1

3. Secondary Outcome: Progression-free Survival
Description: Proportion of patients alive without progression 1 year from the start of study therapy
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

4. Secondary Outcome: Proportion of Patients Undergoing Surgery
Description: Proportion of patients who underwent surgical resection after receiving neoadjuvant therapy
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

5. Secondary Outcome: Overall Survival
Description: Overall survival 1 year after the initiation of study therapy
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

6. Secondary Outcome: Proportion of Margin Negative Surgical Resections
Description: Proportion of patients undergoing surgical resection with surgical margins uninvolved by tumor
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 2 | 1
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 18 months
Description: Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=2) | Arm B (N=1)
Hematoma Grade 3 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nausea Grade 3 (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain Grade 3 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anorexia Grade 3 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=2) | Arm B (N=1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Thrush (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fatigue (Nervous system disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Cellulitis left arm (Infections and infestations) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bartholin's gland cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT03519308/Prot_SAP_000.pdf